CLINICAL TRIAL: NCT05966324
Title: A Phase 1 Single and Multiple Dose Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of Baxdrostat in Healthy Japanese and Caucasian Subjects
Brief Title: Baxdrostat Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study in a Japanese Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIN-107-126
Record Dates: First submitted 2023-07-04; First posted 2023-07-28 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hypertension
Keywords: hypertension; Japanese; PK; baxdrostat
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This was a single and multiple oral dose study of the safety/tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) in healthy Japanese subjects compared with a cohort of healthy Caucasian subjects. total of 41 subjects were enrolled in this study: 31 Japanese subjects and 10 Caucasian subjects. The study included 4 cohorts and each cohort consisted of 10 subjects, randomized 4:1 (active:placebo). The Japanese cohorts (Cohorts 1, 2, and 4) were performed in parallel. The Caucasian cohort (Cohort 3) was performed after Cohort 2 was complete so that the Caucasian subjects could be matched by certain demographic factors.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study included 4 cohorts and each cohort consisted of 10 subjects, randomized 4:1 (active:placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Oral tablet dose of baxdrostat 1 mg or placebo, administered as a single dose (Day 1) and multiple doses (once daily [QD] for 5 days, Days 6 - 10) to Japanese subjects
  Interventions: Drug: baxdrostat
- Cohort 2 (Experimental): Oral tablet dose of baxdrostat 3 mg or placebo, administered as a single dose (Day 1) and multiple doses (QD for 5 days, Days 6 - 10) to Japanese subjects
  Interventions: Drug: baxdrostat
- Cohort 3 (Experimental): Oral tablet dose of baxdrostat 3 mg or placebo, administered as a single dose (Day 1) and multiple doses (QD for 5 days, Days 6 - 10) to Caucasian subjects
  Interventions: Drug: baxdrostat
- Cohort 4 (Experimental): Oral tablet dose of baxdrostat 10 mg or placebo, administered as a single dose (Day 1) and multiple doses (QD for 5 days, Days 6 - 10) to Japanese subjects
  Interventions: Drug: baxdrostat

INTERVENTIONS:
Drug: baxdrostat — Baxdrostat is an aldosterone synthase inhibitor
  Other Names: CIN-107

SUMMARY:
The goal of this study is to compare the characteristics of baxdrostat (CIN-107) in terms of baxdrostat levels over time in the blood in healthy Japanese and Caucasian volunteer participants.

DETAILED DESCRIPTION:
Main Objectives were:

* To assess the safety and tolerability of single and multiple oral doses of baxdrostat in healthy Japanese subjects.
* To assess pharmacokinetics (PK) of baxdrostat and CIN-107-M after single and multiple oral doses of baxdrostat in healthy Japanese subjects.
* To assess pharmacodynamic (PD) effects of single and multiple oral doses of baxdrostat in healthy Japanese subjects.
* To compare the PK and PD of baxdrostat and CIN-107-M after single and multiple oral doses of baxdrostat between Japanese and Caucasian subjects.

Participants will take baxdrostat and have their safety and blood levels of baxdrostat measured over several days following single and multiple dose administration of 3 different dose levels of baxdrostat. The baxdrostat blood levels over time and the levels of certain hormones that regulate blood pressure will be compared between the dose groups and between the healthy Japanese and Caucasian volunteer participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 to 55 years of age, inclusive.
* Demographics as follows:

  1. Japanese subjects must have been born in Japan, with both biological parents and all 4 biological grandparents of Japanese descent, have lived outside of Japan for < 10 years, and have not significantly changed his or her diet since leaving Japan (eg, still mainly eating a "Japanese" diet), OR
  2. Caucasian ancestry (Cohort 3)
* Healthy status as defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, and laboratory assessments (hematology, chemistry, serology, and urinalysis).
* A BMI between 18 - 30 kg/m2, inclusive.
* Females may be of nonchildbearing or childbearing potential. Females of nonchildbearing potential are postmenopausal or surgically sterile. Females of nonchildbearing potential are exempt from the dual contraception requirement.

Females of childbearing potential may be included, provided the subject agrees to continuously use dual methods of contraception from 1 month prior through 90 days after study drug administration.

* Able to participate and willing to give written informed consent and to comply with the study restrictions.

Exclusion Criteria:

1. Any clinically relevant history or the presence of respiratory, renal, hepatic, gastrointestinal, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, allergic, ophthalmological disease or connective tissue disease, cancer or cirrhosis.
2. A history of clinically significant drug hypersensitivity.
3. Subjects with clinically significant symptoms of an infectious illness (bacterial, viral, or parasitic) within 5 days of the first dose or a history of recurrent infections.
4. History of alcohol abuse, illicit drug use, physical dependence to any opioid, or any history of drug abuse or addiction (including soft drugs like cannabis products) within 6 months of screening.
5. Nicotine users unable or unwilling to restrict nicotine usage to the equivalent of 5 cigarettes daily during the study and to not smoke during the in-clinic stays. (Nicotine-containing products include cigarettes, chewing tobacco, snuff, nicotine patches, electronic cigarettes, vaping devices, etc.)
6. Positive result for HIV-1 or HIV-2, hepatitis C virus (HCV), or HBsAg at screening.
7. Confirmed (based on the average of ≥ 3 blood pressure measurements) sustained systolic blood pressure > 140 or < 90 mmHg, and diastolic blood pressure > 90 or < 45 mmHg, and pulse rate > 100 or < 40 bpm.
8. Personal or family history of congenital long QT syndrome or QTcF values > 450 msec in males or > 470 msec in females.
9. Screening or baseline ECGs with QRS and/or T-wave judged by the Investigator to be unfavorable for a consistently accurate QT measurement (ie, neuromuscular artifact that cannot be readily eliminated, arrhythmias, indistinct QRS onset, low amplitude T-wave, merged T- and U-waves, prominent U-waves, etc.)
10. Screening or baseline ECG with clinically significant abnormalities such as atrial fibrillation, atrial flutter, complete bundle branch block, Wolf-Parkinson-White Syndrome, or cardiac pacemaker, as judged by the Investigator.
11. Clinically significant abnormalities in laboratory test results (including hepatic and renal panels, complete blood count, chemistry panel, and urinalysis) at screening or prior to dosing. The Medical Monitor may be consulted to discuss questionable abnormalities. Laboratory values that are not clinically significant, in the Investigator's opinion, may be allowable. In addition, subjects with the following will be excluded from the study (regardless of significance):

    * red blood cell count < 0.75 x lower limit of normal (LLN)
    * white blood cell count < 0.75 x LLN
    * hemoglobin < 0.75 x LLN
    * aspartate transaminase > 1.25 x upper limit of normal (ULN)
    * alanine aminotransferase > 1.25 x ULN
    * potassium > ULN
    * sodium < LLN

    In case of questionable results, tests performed during screening or Day -2 may be repeated before dosing to confirm eligibility.
12. Subjects with estimated glomerular filtration rate < 60 mL/min (according to the Modification of Diet in Renal Disease formula).
13. Subjects with clinically significant orthostatic hypotension (defined as a decrease in systolic blood pressure of ≥ 20 mmHg or a decrease in diastolic blood pressure of ≥ 10 mmHg at 2 minutes of standing).
14. Donation of blood > 450 mL within 3 months prior to screening or plasma within 14 days of dose administration.
15. Concomitant disease or condition that could interfere with, or for which the treatment thereof, might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this study.
16. Known intolerance to cosyntropin test product.
17. Use of prescription, over-the-counter, or herbal medications within 14 days prior to dose administration.
18. Participation in an investigational drug or device study within 30 days or 5 half-lives, whichever is longer, prior to dosing.
19. Corticosteroid use (systemic or extensive topical use) within 3 months prior to dosing.
20. Has received a vaccination within 14 days prior to administration of the study drug.
21. Males must agree to not donate sperm from screening through 90 days after study drug administration has been completed.
22. Strenuous activity (as assessed by the Investigator) within 48 hours prior to clinical site admission.
23. Consumption of alcohol or caffeine-containing food or beverages within 3 days prior to admission to the clinical site.
24. Involved in the planning or conduct of this study.
25. Unwilling or unlikely to comply with the requirements of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events following single and multiple doses of baxdrostat in healthy Japanese and Caucasian participants versus placebo recipients. | 0 to 19 days after dosing
  Safety and tolerability will be assessed by comparison of number of treatment emergent adverse events between groups.
Area under the curve (AUC) for baxdrostat and the CIN-107-M metabolite after single and multiple oral doses of baxdrostat in healthy Japanese subjects. | 0 to 15 days after dosing
  AUC [0 to 24 hours, 0 to last quantifiable concentration, and 0 to infinity of baxdrostat] will be determined for baxdrostat and the CIN-107M metabolite for Japanese participants in each of each of the 3 dose groups of baxdrostat.
Maximum Plasma Concentration [Cmax] of baxdrostat and the CIN-107-M metabolite after single and multiple oral doses of baxdrostat in healthy Japanese subjects. | 0 to 15 days after dosing
  Cmax will be determined for baxdrostat and the CIN-107M metabolite for Japanese participants in each of each of the 3 dose groups of baxdrostat.
Plasma aldosterone levels following single and multiple oral doses of baxdrostat in healthy Japanese subjects. | 0 to 15 days after dosing
  Plasma aldosterone levels will be determined for baxdrostat and the CIN-107M metabolite for Japanese participants in each of each of the 3 dose groups of baxdrostat.
Time to Maximum Plasma Concentration [Tmax] of baxdrostat and the CIN-107-M metabolite after single and multiple oral doses of baxdrostat in healthy Japanese subjects. | 0 to 15 days after dosing
  Tmax will be determined for baxdrostat and the CIN-107M metabolite for Japanese participants in each of each of the 3 dose groups of baxdrostat.
Terminal elimination half-life of baxdrostat and the CIN-107-M metabolite after single and multiple oral doses of baxdrostat in healthy Japanese subjects. | 0 to 15 days after dosing
  Terminal elimination half-life will be determined for baxdrostat and the CIN-107M metabolite for Japanese participants in each of each of the 3 dose groups of baxdrostat.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Winkle, MD, Principal Investigator — ICON Clinical Research LLC
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CIN-107-126&attachmentIdentifier=d22fa00b-6fa7-4160-89b5-9b41508786b5&fileName=cin-107-126-synopsis_Redacted.pdf&versionIdentifier=